CLINICAL TRIAL: NCT02971423
Title: A Phase I, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Intravenous ETX2514 Administered in Healthy Subjects
Brief Title: Evaluation of the Safety, Tolerability and Pharmacokinetics of Intravenous ETX2514 Administered in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Entasis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS2514-2016-0001; ACTRN12616000995471p (Registry Identifier: Australian New Zealand Clinical Trials Registry (ANZCTR))
Record Dates: First submitted 2016-10-21; First posted 2016-11-23 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-04

CONDITIONS: Acinetobacter Baumannii Infection
Keywords: infection; gram-negative bacterium
MeSH Terms: conditions — Infections | interventions — durlobactam; Sulbactam; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (15):
- Part A; Cohort 1: 0.25 g IV ETX2514/placebo (Experimental): Part A of the study will explore the safety and tolerability of a single ascending dose (SAD) of intravenous (IV) ETX2514. Participants in Cohort 1, aged 18 to 55 years, will receive 0.25 grams (g) IV ETX2514/placebo infused over 3 hours.
  Interventions: Drug: ETX2514; Drug: Placebo
- Part A; Cohort 2: 0.5 g IV ETX2514/placebo (Experimental): Part A of the study will explore the safety and tolerability of a SAD of IV ETX2514. Participants in Cohort 2, aged 18 to 55 years, will receive 0.5 g IV ETX2514/placebo infused over 3 hours.
  Interventions: Drug: ETX2514; Drug: Placebo
- Part A; Cohort 3: 1.0 g IV ETX2514/placebo (Experimental): Part A of the study will explore the safety and tolerability of a SAD of IV ETX2514. Participants in Cohort 3, aged 18 to 55 years, will receive 1.0 g IV ETX2514/placebo infused over 3 hours.
  Interventions: Drug: ETX2514; Drug: Placebo
- Part A; Cohort 4: 1.0 g IV ETX2514/placebo (Experimental): Part A of the study will explore the safety and tolerability of a SAD of IV ETX2514. Participants in Cohort 4, aged 18 to 55 years, will receive 1.0 g IV ETX2514/placebo infused over 2 hours.
  Interventions: Drug: ETX2514; Drug: Placebo
- Part A; Cohort 5: 2.0 g IV ETX2514/placebo (Experimental): Part A of the study will explore the safety and tolerability of a SAD of IV ETX2514. Participants in Cohort 5, aged 18 to 55 years, will receive 2.0 g IV ETX2514/placebo infused over 3 hours.
  Interventions: Drug: ETX2514; Drug: Placebo
- Part A; Cohort 6: 4.0 g IV ETX2514/placebo (Experimental): Part A of the study will explore the safety and tolerability of a SAD of IV ETX2514. Participants in Cohort 5, aged 18 to 55 years, will receive 4.0 g IV ETX2514/placebo infused over 3 hours.
  Interventions: Drug: ETX2514; Drug: Placebo
- Part A; Cohort 7: 8.0 g IV ETX2514/placebo (Experimental): Part A of the study will explore the safety and tolerability of a SAD of IV ETX2514. Participants in Cohort 7, aged 18 to 55 years, will receive 8.0 g IV ETX2514/placebo infused over 3 hours.
  Interventions: Drug: ETX2514; Drug: Placebo
- Part A; Cohort 8: 1.0 g IV ETX2514/placebo (Experimental): Part A of the study will explore the safety and tolerability of a SAD of IV ETX2514. Participants in Cohort 8, aged 65 years or older, will receive 1.0 g IV ETX2514/placebo infused over 3 hours.
  Interventions: Drug: ETX2514; Drug: Placebo
- Part B; Cohort 9: 0.25 g IV EXT2514/placebo (Experimental): Part B of the study will explore the safety and tolerability of multiple ascending doses (MAD) of IV ETX2514. Participants in Cohort 9, aged 18 to 55 years, will receive 0.25 g IV EXT2514/placebo infused over 3 hours, every 6 hours (4 times a day) for 7 consecutive days, and then will receive 1 dose on Day 8.
  Interventions: Drug: ETX2514; Drug: Placebo
- Part B; Cohort 10: 0.5 g IV EXT2514/placebo (Experimental): Part B of the study will explore the safety and tolerability of MAD of IV ETX2514. Participants in Cohort 10, aged 18 to 55 years, will receive 0.5 g IV EXT2514/placebo infused over 3 hours, every 6 hours (4 times a day) for 7 consecutive days, and then will receive 1 dose on Day 8.
  Interventions: Drug: ETX2514; Drug: Placebo
- Part B; Cohort 11: 1.0 g IV EXT2514/placebo (Experimental): Part B of the study will explore the safety and tolerability of MAD of IV ETX2514. Participants in Cohort 11, aged 18 to 55 years, will receive 1.0 g IV EXT2514/placebo infused over 3 hours, every 6 hours (4 times a day) for 7 consecutive days, and then will receive 1 dose on Day 8.
  Interventions: Drug: ETX2514; Drug: Placebo
- Part B; Cohort 12: 2.0 g IV EXT2514/placebo (Experimental): Part B of the study will explore the safety and tolerability of MAD of IV ETX2514. Participants in Cohort 12, aged 18 to 55 years, will receive 2.0 g IV EXT2514/placebo infused over 3 hours, every 6 hours (4 times a day) for 7 consecutive days, and then will receive 1 dose on Day 8.
  Interventions: Drug: ETX2514; Drug: Placebo
- Part C; Cohort 13: ETX2514/placebo with sulbactam (Experimental): Part C of the study will explore the safety and tolerability of IV ETX2514 when administered as a single dose in combination with sulbactam (1.0 g) and/or imipenem/cilastatin (0.5 g) to healthy participants. On Day 1, participants will receive a single dose of 1.0 g IV ETX2514/placebo infused over 3 hours. On Day 3, participants will receive a single dose of 1.0 g IV sulbactam infused over 3 hours. On Day 5, participants will receive a single dose of 1.0 g IV ETX2514/placebo plus 1.0 g sulbactam infused over 3 hours at the same time. The actual Day 1 and Day 5 ETX2514 dose and infusion time will be determined based on PK and safety data from Part A.
  Interventions: Drug: ETX2514; Drug: Placebo; Drug: Sulbactam
- Part C; Cohort 14: ETX2514/placebo with SUL and/or IM/CIL (Experimental): Part C of the study will explore the safety and tolerability of IV ETX2514 when administered as a single dose in combination with sulbactam (SUL: 1.0 g) and/or imipenem/cilastatin (IM/CIL: 0.5 g) to healthy participants. On Day 1, participants will receive a single dose of 1.0 g IV ETX2514/placebo infused over 3 hours. On Day 3, participants will receive a single dose of 0.5 g IV imipenem/cilastatin infused over 30 minutes. On Day 5, participants will receive a single dose of 1.0 g IV ETX2514/placebo infused over 3 hours plus 0.5 g imipenem/cilastatin infused over 30 minutes initiated at the same time as ETX2514/placebo. On Day 8, participants will receive a single dose of 1.0 g IV ETX2514/placebo plus 1.0 g sulbactam infused over 3 hours at the same time plus 0.5 g imipenem/cilastatin infused over 30 minutes initiated at the same time as ETX2514/placebo. The actual Day 1, Day 5, and Day 8 ETX2514 dose and infusion time will be determined based on PK and safety data from Part A.
  Interventions: Drug: ETX2514; Drug: Placebo; Drug: Sulbactam; Drug: Imipenem/Cilastatin
- Part D; Cohort 15: ETX2514/placebo with SUL and/or IM/CIL (Experimental): Part D of the study will explore the safety and tolerability of multiple doses of combined IV ETX2514/sulbactam (1.0 g)/imipenem/cilastatin (0.5 g) to healthy participants. Participants in Cohort 15 will receive 1.0 g IV ETX2514/placebo and 1.0 g IV sulbactam both infused over 3 hours and 0.5 g IV imipenem/cilastatin infused over 30 minutes every 6 hours (4 times a day) for 10 days and will receive 1 dose on Day 11. The actual ETX2514 dose and infusion time will be determined based on PK and safety data from Part C.
  Interventions: Drug: ETX2514; Drug: Placebo; Drug: Sulbactam; Drug: Imipenem/Cilastatin

INTERVENTIONS:
Drug: ETX2514
Drug: Placebo — matching placebo infusion
Drug: Sulbactam
  Arms: Part C; Cohort 13: ETX2514/placebo with sulbactam; Part C; Cohort 14: ETX2514/placebo with SUL and/or IM/CIL; Part D; Cohort 15: ETX2514/placebo with SUL and/or IM/CIL
Drug: Imipenem/Cilastatin
  Arms: Part C; Cohort 14: ETX2514/placebo with SUL and/or IM/CIL; Part D; Cohort 15: ETX2514/placebo with SUL and/or IM/CIL

SUMMARY:
This research project is being conducted to look at the safety, tolerability, and pharmacokinetics (PK; how the human body processes a substance) of ETX2514 when given to healthy volunteers intravenously as a single dose, and when given as multiple intravenous doses for up to 8 consecutive days.

As it is anticipated that ETX2514 could be used as a treatment for Acinetobacter baumannii (a type of bacteria) infections, this project will also look at whether ETX2514 will interact with the current treatments for these infections when they are administered at the same time.

DETAILED DESCRIPTION:
This Phase 1, single-center, randomized, double-blind, and placebo-controlled study investigates the safety, tolerability, and PK profile of single and multiple ascending doses of intravenous (IV) ETX2514 when administered intravenously alone and in combination with sulbactam and/or imipenem/cilastatin in healthy adult participants.

The study will be conducted in four Parts: A, B, C, and D. Part A will explore the safety and tolerability of a single ascending dose (SAD) of IV ETX2514 over 8 cohorts. Part B will explore the safety and tolerability of multiple ascending doses (MAD) of IV ETX2514 over 4 cohorts. Part C will explore the safety and tolerability of IV ETX2514 when administered as a single dose in combination with sulbactam (1.0 gram [g]) and/or imipenem/cilastatin (0.5 g) to healthy participants over 2 cohorts. Part D will explore the safety and tolerability of multiple doses of combined IV ETX2514/sulbactam (1.0 g)/imipenem/cilastatin (0.5 g) to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 55 years (inclusive). In addition, 8 participants greater than or equal to 65 years of age will be enrolled.
* Be in general good health without a clinically significant medical history
* Provide voluntary written informed consent prior to any study procedures and are willing and able to comply with the prescribed treatment protocol and evaluations
* Body mass index (BMI) greater than or equal to 18.0 kilograms (kg)/meters square (m^2) and less than or equal to 32.0 kg/m^2
* Clinical laboratory values within the normal limits as defined by the clinical laboratory, unless the Principal Investigator decides that out-of-range values are not clinically significant
* Negative screen for drugs of abuse, alcohol, hepatitis B surface antigen (HBS Ag), hepatitis C virus antibody (HCV Ab), and Human Immunodeficiency Virus (HIV) at screening; and drugs of abuse, alcohol pre dose on Day -1
* Female participants must be of non-childbearing potential, or using a medically acceptable contraceptive regimen and must have a negative pregnancy test at Screening (serum) and on Day -1 (urine) prior to study drug dosing. Male participants must be surgically sterile, or using a medically acceptable contraceptive regimen.

Exclusion Criteria:

* History of any moderate or severe hypersensitivity or allergic reaction to any beta-lactam antimicrobial (e.g., penicillin, cephalosporin, sulbactam, or carbapenem).
* Use of prescription or over the counter medications within 7 days of Investigational Product administration, with the exception of contraceptive medications, paracetamol, oral non-steroidal anti-inflammatory agents, topical over the counter preparations, and routine vitamins (if they do not exceed an intake of 20 to 600 times the recommended daily dose), unless agreed as non-clinically relevant by the Principal Investigator and Sponsor
* Participation in an investigational drug or device study within 30 days before study drug dosing, i.e., there was at least 30 days in between the last dose on a prior study and dose administration on this study
* Current smoker, or difficulty abstaining from smoking for the duration of study confinement
* History of major organ dysfunction
* Infection or any serious underlying medical condition that would impair the participant from receiving study drug
* History of excessive alcohol intake (more than 4 standard drinks daily, on average) or use of recreational drugs within the last 3 months
* Standard donation of blood within 30 days of the study
* Concomitant disease or condition, including laboratory abnormality, which could interfere with the conduct of the study, or which would, in the opinion of the investigator, pose an unacceptable risk to the participant in this study
* Anticipated need for surgery or hospitalization during the study
* Unwillingness or inability to comply with the study protocol for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with any non-serious and any serious adverse event | up to 14 days after the last infusion of study drug (Study Day 182)
Number of participants with an adverse event of the indicated causality and severity | up to 14 days after the last infusion of study drug (Study Day 182)
Number of participants with abnormal, clinically significant hematology and clinical chemistry laboratory values at the indicated time points in Part A | Baseline (Day -1); Days 3, 5, 7, and 15 (Follow-up)
Number of participants with abnormal, clinically significant hematology and clinical chemistry laboratory values at the indicated time points in Part B | Baseline (Day -1; Study Day [SD] 37); Days 2, 3, 5, 7, and 10 (SDs 39, 40, 42, 44, and 47, respectively); Day 22 (SD 59; Follow-up)
Number of participants with abnormal, clinically significant hematology and clinical chemistry laboratory values at the indicated time points in Part C | Cohort 13: Baseline (Day -1; Study Day [SD] 80); Days 3, 4, and 7 (SDs 83, 84, and 87, respectively); Day 19 (SD 99; Follow-up). Cohort 14: Baseline; Days 3, 4, 7, and 10 (SDs 83, 84, 87, and 90, respectively); Day 22 (SD 102; Follow-up)
Number of participants with abnormal, clinically significant hematology and clinical chemistry laboratory values at the indicated time points in Part D | Baseline (Day -1; SD 122); Days 2, 3, 5, 7, 10, 11, and 13 (SDs 124, 125, 127, 129, 132, and 133, respectively); Day 25 (SD 147; Follow-up)
Change from Baseline in vital signs at the indicated time points in Part A | Baseline (Day -1); Days 1-3; Day 5; Day 7; Day 15 (Follow-up)
  Day 1: prior to infusion, and 1, 3, 6, and 12 hours post start of infusion. Day 2: 24 hours post start of infusion). Day 3: 48 hours post start of infusion
Change from Baseline in vital signs at the indicated time points in Part B | Baseline (Day -1; SD 37); Days 1-10 (SDs 38-47, respectively); Day 22 (SD 59; Follow-up)
  Days 1-8: 30 minutes prior to infusion and 3, 6, and 12 hours post start of infusion. Day 9: 24 hours post Day 8 start of infusion. Day 10: 48 hours post Day 8 start of infusion
Change from Baseline in vital signs at the indicated time points in Cohort 13 of Part C | Baseline (Day -1; SD 80); Days 1-7 (SDs 81-87, respectively); Day 19 (SD 99; Follow-up)
  Days 1, 3, and 5: 30 minutes prior to infusion and 3, 6, and 12 hours post start of infusion. Days 2, 4, and 6: 24 hours post start of infusion. Day 7: 48 hours post Day 5 start of infusion
Change from Baseline in vital signs at the indicated time points in Cohort 14 of Part C | Baseline (Day -1; SD 80); Days 1-10 (SDs 81-90, respectively); Day 22 (SD 102; Follow-up)
  Days 1, 3, 5, and 8: 30 minutes prior to infusion and 3, 6, and 12 hours post start of infusion. Days 2, 4, 6, and 9: 24 hours post start of infusion. Days 7 and 10: 48 hours post Day 5 and Day 8, respectively, start of infusion
Change from Baseline in vital signs at the indicated time points in Part D | Baseline (SD 122); Days 1-13 (SDs 123-135, respectively); Day 25 (SD 147; Follow-up)
  Days 1-11: 30 minutes prior to infusion and 3, 6, and 12 hours post infusion
Change from Baseline in electrocardiogram parameters at the indicated time points in Parts A and B | Part A: Baseline (Day -1); Days 1 and 3; Follow-up visit (Day 15). Part B: Baseline (Day -1; SD 37); Days 1, 3, 5, 7, 10, and 22 (SDs 38, 40, 42, 44, 47, and 59, respectively)
  Part A: Day 1: 150 minutes after start of infusion; Day 3: 48 hours after start of infusion. Part B: Days 1, 3, 5, and 7: 150 minutes after start of infusion; Day 10: 48 hours post Day 8 start of infusion
Change from Baseline in electrocardiogram parameters at the indicated time points in Cohort 13 in Part C | Baseline (Day -1; SD 80); Days 1, 3, 5, and 7 (SDs 81, 83, 85, and 87, respectively); Day 19 (SD 99; Follow-up)
  Days 1, 3, and 5: 150 minutes post start of infusion; Day 7: 48 hours post Day 5 start of infusion
Change from Baseline in electrocardiogram parameters at the indicated time points in Cohort 14 in Part C | Baseline (Day -1; SD 80); Days 1, 3, 5, 8, and 10 (SDs 81, 83, 85, 88, and 90, respectively); Day 22 (SD 102; Follow-up)
  Days 1, 3, 5, and 8: 150 minutes post start of infusion; Day 10: 48 hours post Day 8 start of infusion
Change from Baseline in electrocardiogram parameters at the indicated time points in Part D | Baseline (SD 122); Days 1, 3, 5, 7, 9, and 11 (SDs 123, 125, 127, 129, 131, and 133, respectively); Day 13 (SD 135); Day 25 (SD 147; Follow-up)
  Days 1, 3, 5, 7, 9, and 11: 150 minutes post start of infusion. Day 13: 48 hours post Day 11 start of infusion
Number of participants with an infusion site reaction | up to 14 days after the last infusion of study drug (SD 182)
Mean peak plasma concentration (Cmax) and plasma concentration at time t (Ct) in blood at the indicated time points in Cohorts 1-3 and 5-8 in Part A | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean Cmax and Ct in blood at the indicated time points in Cohort 4 in Part A | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 2.5, 3, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean Cmax and Ct in blood at the indicated time points in Part B | Days 1, 2, 4, 8, 9, and 10 (SDs 38, 39, 41, 45, 46, and 47, respectively)
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 8: 30 minutes prior to infusion of the final dose, which is given on Day 8; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 9: 24 and 36 hours post start of infusion. Day 10: 48 hours post start of infusion
Mean Cmax and Ct in blood at the indicated time points in Cohort 13 in Part C | Days 1-7 (SDs 81-87, respectively)
  Day 1: 30 minutes prior to infusion of ETX2514/placebo; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of ETX2514/placebo. Day 2: 24 and 36 hours post start of infusion of ETX2514/placebo. Day 3: immediately prior to start of infusion of sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of sulbactam. Day 4: 24 and 36 hours post start of infusion of sulbactam. Day 5: immediately prior to infusion to co-administer ETX2514/placebo and sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 6: 24 and 36 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 7: 48 hours post start of infusion to co-administer ETX2514/placebo and sulbactam
Mean Cmax and Ct in blood at the indicated time points in Cohort 14 in Part C | Days 1-10 (SDs 81-90, respectively)
  ETX2514/placebo infusion: Day 1: 30 minutes prior to infusion (PTI); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion (PSOI). Day 2: 24 and 36 PSOI. Imipenem (IM)/cilastatin (CIL) infusion: Day 3: immediately prior to start of infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 4, 5, 6, 8, and 12 hours PSOI. Day 4: 24 and 36 hours PSOI. Co-administration of ETX2514/placebo and IM/CIL: Day 5: immediately prior to infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours PSOI. Day 6: 24 and 36 hours PSOI. Day 7: 48 hours PSOI. Co-administration of ETX2514/placebo, sulbactam, and IM/CIL: Day 8: 30 minutes prior to infusion; 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 PSOI. Day 9: 24 and 36 hours PSOI. Day 10: 48 hours PSOI
Mean Cmax and Ct in blood at the indicated time points in Part D | Days 1, 2, 4, 11, 12, and 13 (SDs 124, 125, 127, 134, 135, and 136, respectively)
  Day 1: 30 minutes prior to infusion; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 11: 30 minutes prior to infusion of the final dose given on Day 11; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 12: 24 and 36 hours post start of infusion. Day 13: 48 hours post start of infusion
Mean time to peak plasma concentration (Tmax) in blood at the indicated time points in Cohorts 1-3 and 5-8 in Part A | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean Tmax in blood at the indicated time points in Cohort 4 in Part A | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 2.5, 3, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean Tmax in blood at the indicated time points in Part B | Days 1, 2, 4, 8, 9, and 10 (SDs 38, 39, 41, 45, 46, and 47, respectively)
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 8: 30 minutes prior to infusion of the final dose, which is given on Day 8; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 9: 24 and 36 hours post start of infusion. Day 10: 48 hours post start of infusion
Mean Tmax in blood at the indicated time points in Cohort 13 in Part C | Days 1-7 (SDs 81-87, respectively)
  Day 1: 30 minutes prior to infusion of ETX2514/placebo; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of ETX2514/placebo. Day 2: 24 and 36 hours post start of infusion of ETX2514/placebo. Day 3: immediately prior to start of infusion of sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of sulbactam. Day 4: 24 and 36 hours post start of infusion of sulbactam. Day 5: immediately prior to infusion to co-administer ETX2514/placebo and sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 6: 24 and 36 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 7: 48 hours post start of infusion to co-administer ETX2514/placebo and sulbactam
Mean Tmax in blood at the indicated time points in Cohort 14 in Part C | Days 1-10 (SDs 81-90, respectively)
  ETX2514/placebo infusion: Day 1: 30 minutes prior to infusion (PTI); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion (PSOI). Day 2: 24 and 36 PSOI. Imipenem (IM)/cilastatin (CIL) infusion: Day 3: immediately prior to start of infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 4, 5, 6, 8, and 12 hours PSOI. Day 4: 24 and 36 hours PSOI. Co-administration of ETX2514/placebo and IM/CIL: Day 5: immediately prior to infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours PSOI. Day 6: 24 and 36 hours PSOI. Day 7: 48 hours PSOI. Co-administration of ETX2514/placebo, sulbactam, and IM/CIL: Day 8: 30 minutes prior to infusion; 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 PSOI. Day 9: 24 and 36 hours PSOI. Day 10: 48 hours PSOI
Mean Tmax in blood at the indicated time points in Part D | Days 1, 2, 4, 11, 12, and 13 (SDs 124, 125, 127, 134, 135, and 136, respectively)
  Day 1: 30 minutes prior to infusion; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 11: 30 minutes prior to infusion of the final dose given on Day 11; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 12: 24 and 36 hours post start of infusion. Day 13: 48 hours post start of infusion
Mean AUC from time 0 to 24 hours (AUC0-24), AUC from time 0 to the last time point evaluated (AUC0-t), and AUC from time 0 and extrapolated to infinity (AUC0-∞) in blood at the indicated time points in Cohorts 1-3 in Part A | Days 1-3
  AUC is defined as area under the concentration time curve. Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean AUC0-24, AUC0-t, and AUC0-∞ in blood at the indicated time points in Cohort 4 in Part A | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 2.5, 3, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean AUC0-24, AUC0-t, and AUC0-∞ in blood at the indicated time points in Part B | Days 1, 2, 4, 8, 9, and 10 (SDs 38, 39, 41, 45, 46, and 47, respectively)
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 8: 30 minutes prior to infusion of the final dose, which is given on Day 8; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 9: 24 and 36 hours post start of infusion. Day 10: 48 hours post start of infusion
Mean AUC0-24, AUC0-t, and AUC0-∞ in blood at the indicated time points in Cohort 13 in Part C | Days 1-7 (SDs 81-87, respectively)
  Day 1: 30 minutes prior to infusion of ETX2514/placebo; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of ETX2514/placebo. Day 2: 24 and 36 hours post start of infusion of ETX2514/placebo. Day 3: immediately prior to start of infusion of sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of sulbactam. Day 4: 24 and 36 hours post start of infusion of sulbactam. Day 5: immediately prior to infusion to co-administer ETX2514/placebo and sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 6: 24 and 36 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 7: 48 hours post start of infusion to co-administer ETX2514/placebo and sulbactam
Mean AUC0-24, AUC0-t, and AUC0-∞ in blood at the indicated time points in Cohort 14 in Part C | Days 1-10 (SDs 81-90, respectively)
  ETX2514/placebo infusion: Day 1: 30 minutes prior to infusion (PTI); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion (PSOI). Day 2: 24 and 36 PSOI. Imipenem (IM)/cilastatin (CIL) infusion: Day 3: immediately prior to start of infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 4, 5, 6, 8, and 12 hours PSOI. Day 4: 24 and 36 hours PSOI. Co-administration of ETX2514/placebo and IM/CIL: Day 5: immediately prior to infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours PSOI. Day 6: 24 and 36 hours PSOI. Day 7: 48 hours PSOI. Co-administration of ETX2514/placebo, sulbactam, and IM/CIL: Day 8: 30 minutes prior to infusion; 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 PSOI. Day 9: 24 and 36 hours PSOI. Day 10: 48 hours PSOI
Mean AUC0-24, AUC0-t, and AUC0-∞ in blood at the indicated time points in Part D | Days 1, 2, 4, 11, 12, and 13 (SDs 124, 125, 127, 134, 135, and 136, respectively)
  Day 1: 30 minutes prior to infusion; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 11: 30 minutes prior to infusion of the final dose given on Day 11; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 12: 24 and 36 hours post start of infusion. Day 13: 48 hours post start of infusion
Mean elimination rate constant (Kel) in blood at the indicated time points in Cohorts 1-3 and 5-8 in Part A | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean Kel in blood at the indicated time points in Cohort 4 in Part A | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 2.5, 3, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean Kel in blood at the indicated time points in Part B | Days 1, 2, 4, 8, 9, and 10 (SDs 38, 39, 41, 45, 46, and 47, respectively)
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 8: 30 minutes prior to infusion of the final dose, which is given on Day 8; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 9: 24 and 36 hours post start of infusion. Day 10: 48 hours post start of infusion
Mean Kel in blood at the indicated time points in Cohort 13 in Part C | Days 1-7 (SDs 81-87, respectively)
  Day 1: 30 minutes prior to infusion of ETX2514/placebo; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of ETX2514/placebo. Day 2: 24 and 36 hours post start of infusion of ETX2514/placebo. Day 3: immediately prior to start of infusion of sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of sulbactam. Day 4: 24 and 36 hours post start of infusion of sulbactam. Day 5: immediately prior to infusion to co-administer ETX2514/placebo and sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 6: 24 and 36 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 7: 48 hours post start of infusion to co-administer ETX2514/placebo and sulbactam
Mean Kel in blood at the indicated time points in Cohort 14 in Part C | Days 1-10 (SDs 81-90, respectively)
  ETX2514/placebo infusion: Day 1: 30 minutes prior to infusion (PTI); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion (PSOI). Day 2: 24 and 36 PSOI. Imipenem (IM)/cilastatin (CIL) infusion: Day 3: immediately prior to start of infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 4, 5, 6, 8, and 12 hours PSOI. Day 4: 24 and 36 hours PSOI. Co-administration of ETX2514/placebo and IM/CIL: Day 5: immediately prior to infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours PSOI. Day 6: 24 and 36 hours PSOI. Day 7: 48 hours PSOI. Co-administration of ETX2514/placebo, sulbactam, and IM/CIL: Day 8: 30 minutes prior to infusion; 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 PSOI. Day 9: 24 and 36 hours PSOI. Day 10: 48 hours PSOI
Mean Kel in blood at the indicated time points in Part D | Days 1, 2, 4, 11, 12, and 13 (SDs 124, 125, 127, 134, 135, and 136, respectively)
  Day 1: 30 minutes prior to infusion; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 11: 30 minutes prior to infusion of the final dose given on Day 11; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 12: 24 and 36 hours post start of infusion. Day 13: 48 hours post start of infusion
Mean elimination half-life (t1/2) in blood at the indicated time points in Cohorts 1-3 and 5-8 in Part A | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean t1/2 in blood at the indicated time points in Cohort 4 in Part A | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 2.5, 3, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean t1/2 in blood at the indicated time points in Part B | Days 1, 2, 4, 8, 9, and 10 (SDs 38, 39, 41, 45, 46, and 47, respectively)
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 8: 30 minutes prior to infusion of the final dose, which is given on Day 8; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 9: 24 and 36 hours post start of infusion. Day 10: 48 hours post start of infusion
Mean t1/2 in blood at the indicated time points in Cohort 13 in Part C | Days 1-7 (SDs 81-87, respectively)
  Day 1: 30 minutes prior to infusion of ETX2514/placebo; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of ETX2514/placebo. Day 2: 24 and 36 hours post start of infusion of ETX2514/placebo. Day 3: immediately prior to start of infusion of sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of sulbactam. Day 4: 24 and 36 hours post start of infusion of sulbactam. Day 5: immediately prior to infusion to co-administer ETX2514/placebo and sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 6: 24 and 36 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 7: 48 hours post start of infusion to co-administer ETX2514/placebo and sulbactam
Mean t1/2 in blood at the indicated time points in Cohort 14 in Part C | Days 1-10 (SDs 81-90, respectively)
  ETX2514/placebo infusion: Day 1: 30 minutes prior to infusion (PTI); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion (PSOI). Day 2: 24 and 36 PSOI. Imipenem (IM)/cilastatin (CIL) infusion: Day 3: immediately prior to start of infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 4, 5, 6, 8, and 12 hours PSOI. Day 4: 24 and 36 hours PSOI. Co-administration of ETX2514/placebo and IM/CIL: Day 5: immediately prior to infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours PSOI. Day 6: 24 and 36 hours PSOI. Day 7: 48 hours PSOI. Co-administration of ETX2514/placebo, sulbactam, and IM/CIL: Day 8: 30 minutes prior to infusion; 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 PSOI. Day 9: 24 and 36 hours PSOI. Day 10: 48 hours PSOI
Mean t1/2 in blood at the indicated time points in Part D | Days 1, 2, 4, 11, 12, and 13 (SDs 124, 125, 127, 134, 135, and 136, respectively)
  Day 1: 30 minutes prior to infusion; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 11: 30 minutes prior to infusion of the final dose given on Day 11; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 12: 24 and 36 hours post start of infusion. Day 13: 48 hours post start of infusion
Mean clearance in blood at the indicated time points in Cohorts 1-3 and 5-8 in Part A | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean clearance in blood at the indicated time points in Cohort 4 in Part A | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 2.5, 3, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean clearance in urine at the indicated time points in Part A | Baseline (Day -1); Days 1-3
  -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion
Mean clearance in blood at the indicated time points in Part B | Days 1, 2, 4, 8, 9, and 10 (SDs 38, 39, 41, 45, 46, and 47, respectively)
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 8: 30 minutes prior to infusion of the final dose, which is given on Day 8; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 9: 24 and 36 hours post start of infusion. Day 10: 48 hours post start of infusion
Mean clearance in urine at the indicated time points in Part B | Baseline (Day -1; SD 37); Days 1-3 and 7-10 (SDs 38-40 and 44-47, respectively)
  All days: -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion
Mean clearance in blood at the indicated time points in Cohort 13 in Part C | Days 1-7 (SDs 81-87, respectively)
  Day 1: 30 minutes prior to infusion of ETX2514/placebo; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of ETX2514/placebo. Day 2: 24 and 36 hours post start of infusion of ETX2514/placebo. Day 3: immediately prior to start of infusion of sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of sulbactam. Day 4: 24 and 36 hours post start of infusion of sulbactam. Day 5: immediately prior to infusion to co-administer ETX2514/placebo and sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 6: 24 and 36 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 7: 48 hours post start of infusion to co-administer ETX2514/placebo and sulbactam
Mean clearance in urine at the indicated time points in Cohort 13 in Part C | Baseline (Day -1; SD 80); Days 1-7 (SDs 81-87, respectively)
  Day 1 to Day 3 (ETX2514/placebo): from -12 to 0 hours prior to start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion. Days 3-5 (sulbactam): 0-6, 6-12, 12-24, and 24-48 hours post start of infusion. Days 5-7 (infusion to co-administer ETX2514/placebo and sulbactam): 0-6, 6-12, 12-24, and 24-48 hours post start of infusion
Mean clearance in blood at the indicated time points in Cohort 14 in Part C | Days 1-10 (SDs 81-90, respectively)
  ETX2514/placebo infusion: Day 1: 30 minutes prior to infusion (PTI); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion (PSOI). Day 2: 24 and 36 PSOI. Imipenem (IM)/cilastatin (CIL) infusion: Day 3: immediately prior to start of infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 4, 5, 6, 8, and 12 hours PSOI. Day 4: 24 and 36 hours PSOI. Co-administration of ETX2514/placebo and IM/CIL: Day 5: immediately prior to infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours PSOI. Day 6: 24 and 36 hours PSOI. Day 7: 48 hours PSOI. Co-administration of ETX2514/placebo, sulbactam, and IM/CIL: Day 8: 30 minutes prior to infusion; 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 PSOI. Day 9: 24 and 36 hours PSOI. Day 10: 48 hours PSOI
Mean clearance in urine at the indicated time points in Cohort 14 in Part C | Baseline (Day -1; SD 80); Days 1-10 (SDs 81-90, respectively)
  Day 1 to Day 3 (ETX2514/placebo): from -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion. Day 3 to Day 5 (imipenem/cilastatin): 0-6, 6-12, 12-24, and 24-48 hours post start of infusion. Day 5 to Day 7 (infusion to co-administer ETX2514/placebo and imipenem/cilastatin): 0-6, 6-12, 12-24, and 24-48 hours post start of infusion. Day 8 to Day 10 (infusion to co-administer ETX2514/placebo, sulbactam, and imipenem/cilastatin): from -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion
Mean clearance in blood at the indicated time points in Part D | Days 1, 2, 4, 11, 12, and 13 (SDs 124, 125, 127, 134, 135, and 136, respectively)
  Day 1: 30 minutes prior to infusion; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 11: 30 minutes prior to infusion of the final dose given on Day 11; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 12: 24 and 36 hours post start of infusion. Day 13: 48 hours post start of infusion
Mean clearance in urine at the indicated time points in Part D | Baseline (Day -1; SD 123); Days 1-3 (SDs 124-126, respectively); Days 10-13 (SDs 133-136, respectively)
  Days 1-3: from -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion. Days 11-13: from -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion
Mean volume of distribution (VzVdss) in blood at the indicated time points in Cohorts 1-3 and 5-8 in Part A | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean VzVdss in blood at the indicated time points in Cohort 4 in Part A | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 2.5, 3, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean VzVdss in blood at the indicated time points in Part B | Days 1, 2, 4, 8, 9, and 10 (SDs 38, 39, 41, 45, 46, and 47, respectively)
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 8: 30 minutes prior to infusion of the final dose, which is given on Day 8; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 9: 24 and 36 hours post start of infusion. Day 10: 48 hours post start of infusion
Mean VzVdss in blood at the indicated time points in Cohort 13 in Part C | Days 1-7 (SDs 81-87, respectively)
  Day 1: 30 minutes prior to infusion of ETX2514/placebo; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of ETX2514/placebo. Day 2: 24 and 36 hours post start of infusion of ETX2514/placebo. Day 3: immediately prior to start of infusion of sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion of sulbactam. Day 4: 24 and 36 hours post start of infusion of sulbactam. Day 5: immediately prior to infusion to co-administer ETX2514/placebo and sulbactam (48 hours); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 6: 24 and 36 hours post start of infusion to co-administer ETX2514/placebo and sulbactam. Day 7: 48 hours post start of infusion to co-administer ETX2514/placebo and sulbactam
Mean VzVdss in blood at the indicated time points in Cohort 14 in Part C | Days 1-10 (SDs 81-90, respectively)
  ETX2514/placebo infusion: Day 1: 30 minutes prior to infusion (PTI); 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion (PSOI). Day 2: 24 and 36 PSOI. Imipenem (IM)/cilastatin (CIL) infusion: Day 3: immediately prior to start of infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 4, 5, 6, 8, and 12 hours PSOI. Day 4: 24 and 36 hours PSOI. Co-administration of ETX2514/placebo and IM/CIL: Day 5: immediately prior to infusion (48 hours); 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours PSOI. Day 6: 24 and 36 hours PSOI. Day 7: 48 hours PSOI. Co-administration of ETX2514/placebo, sulbactam, and IM/CIL: Day 8: 30 minutes prior to infusion; 30 minutes PSOI; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 PSOI. Day 9: 24 and 36 hours PSOI. Day 10: 48 hours PSOI
Mean VzVdss in blood at the indicated time points in Part D | Days 1, 2, 4, 11, 12, and 13 (SDs 124, 125, 127, 134, 135, and 136, respectively)
  Day 1: 30 minutes prior to infusion; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Days 2 and 4: 30 minutes prior to infusion of the second dose given on Days 2 and 4, respectively. Day 11: 30 minutes prior to infusion of the final dose given on Day 11; 30 minutes post start of infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 12: 24 and 36 hours post start of infusion. Day 13: 48 hours post start of infusion
Mean cumulative excretion of unchanged drug in urine (Ae) at the indicated time points in Part A | Baseline (Day -1); Days 1-3
  -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion
Mean Ae at the indicated time points in Part B | Baseline (Day -1; SD 37); Days 1-3 and 7-10 (SDs 38-40 and 44-47, respectively)
  All days: -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion
Mean Ae at the indicated time points in Cohort 13 in Part C | Baseline (Day -1; SD 80); Days 1-7 (SDs 81-87, respectively)
  Day 1 to Day 3 (ETX2514/placebo): from -12 to 0 hours prior to start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion. Days 3-5 (sulbactam): 0-6, 6-12, 12-24, and 24-48 hours post start of infusion. Days 5-7 (infusion to co-administer ETX2514/placebo and sulbactam): 0-6, 6-12, 12-24, and 24-48 hours post start of infusion
Mean Ae at the indicated time points in Cohort 14 in Part C | Baseline (Day -1; SD 80); Days 1-10 (SDs 81-90, respectively)
  Day 1 to Day 3 (ETX2514/placebo): from -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion. Day 3 to Day 5 (imipenem/cilastatin): 0-6, 6-12, 12-24, and 24-48 hours post start of infusion. Day 5 to Day 7 (infusion to co-administer ETX2514/placebo and imipenem/cilastatin): 0-6, 6-12, 12-24, and 24-48 hours post start of infusion. Day 8 to Day 10 (infusion to co-administer ETX2514/placebo, sulbactam, and imipenem/cilastatin): from -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion
Mean Ae at the indicated time points in Part D | Baseline (Day -1; SD 123); Days 1-3 (SDs 124-126, respectively); Days 10-13 (SDs 133-136, respectively)
  Days 1-3: from -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion. Days 11-13: from -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion

SECONDARY OUTCOMES:
Number of elderly participants with any non-serious and any serious adverse event | up to Day 15
Number of elderly participants with an adverse event of the indicated causality and severity | up to Day 15
Number of participants with abnormal, clinically significant hematology and clinical chemistry parameters at the indicted time points in Part A for elderly participants | Baseline (Day -1); Days 3, 5, 7, and 15 (Follow-up)
Change from Baseline in vital signs at the indicated time points in Part A for elderly participants | Baseline (Day -1); Days 1-3; Day 5; Day 7; Day 15 (Follow-up)
  Day 1: prior to infusion, and 1, 3, 6, and 12 hours post start of infusion. Day 2: 24 hours post start of infusion). Day 3: 48 hours post start of infusion
Change from Baseline in electrocardiogram parameters at the indicated time points in Part A for elderly participants | Baseline (Day -1); Day 1; Day 3; Follow-up visit (Day 15)
  Day 1: 30 minutes after start of infusion
Number of elderly participants with an infusion site reaction | up to Day 15
Mean Cmax and Ct in blood at the indicated time points in Part A for elderly participants | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean Tmax in blood at the indicated time points in Part A for elderly participants | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean AUC0-24, AUC0-t, and AUC0-∞ in blood at the indicated time points in Part A for elderly participants | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean Kel in blood at the indicated time points in Part A for elderly participants | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean t1/2 in blood at the indicated time points in Part A for elderly participants | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean clearance in blood at the indicated time points in Part A for elderly participants | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean clearance in urine at the indicated time points in Part A for elderly participants | Days 1-3
  -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion
Mean VzVdss in blood at the indicated time points in Part A for elderly participants | Days 1-3
  Day 1: 30 minutes prior to infusion; 1, 2, 3, 3.5, 4, 5, 6, 8, and 12 hours post start of infusion. Day 2: 24 and 36 hours post start of infusion; Day 3: 48 hours post start of infusion
Mean Ae at the indicated time points in Part A for elderly participants | Days 1-3
  -12 to 0 hours prior to the start of infusion; 0-6, 6-12, 12-24, and 24-48 hours post start of infusion
Number of elderly participants using concomitant medications | up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, Principal Investigator — Nucleus Network
Locations (1):
- Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Lickliter JD, Lawrence K, O'Donnell J, Isaacs R. Safety, Pharmacokinetics, and Drug-Drug Interaction Potential of Intravenous Durlobactam, a beta-Lactamase Inhibitor, in Healthy Subjects. Antimicrob Agents Chemother. 2020 Jun 23;64(7):e00071-20. doi: 10.1128/AAC.00071-20. Print 2020 Jun 23. PMID 32284380